CLINICAL TRIAL: NCT01358630
Title: Periodontal-, Cardiovascular- and Aneurysmal Diseases.
Brief Title: Vascular and Periodontal Disease - Microbial, Genetic and Histological Causalities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oslo (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Professor, Ph.D., Dr.Odont Ingar Olsen/Professor PhD.MD. Jørgen J. Jørgensen, Institute of Oral Biology, Dental Faculty, University of Oslo/Oslo University Hospital, Departemnt of vascular surgery
Other Study IDs: 08/322b
Record Dates: First submitted 2011-05-19; First posted 2011-05-24 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2010-11

CONDITIONS: Periodontitis; Vascular Disease
Keywords: Periodontitis; Vascular disease; Proinflammatory cytokines
MeSH Terms: conditions — Periodontitis; Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, samples from vascular tissues (atherosclerotic plaques and aneurysmal wall), saliva
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to analyze genetic polymorphisms in genes encoding pro-inflammatory cytokines, and study the genetic predisposition to chronic periodontitis (CP) in combination with atherosclerotic cardiovascular (ACD) and aneurysmal diseases. The investigators will also try to identify oral bacteria in atherosclerotic plaques and aneurysmal walls and thrombus. Histological analyses of atherosclerotic plaques and aneurysmal wall will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing vascular surgery at Oslo University Hospital, Aker, previously randomly collected patients with periodontitis,

Exclusion Criteria:

* patients whom undergone antibiotic treatment the past month.
* patients whom undergone periodontal treatment the past 6 months.
* patients with no teeth

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing vascular surgery at Oslo University Hospital, Aker, previously randomly collected patients with periodontitis, and randomly selected blood donors at Oslo University Hospital, Ullevål.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-10; Primary Completion 2011-03 (Actual); Study Completion 2015-10 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Dental and Medical Faculty, University of Oslo, Oslo, Oslo County, Norway